CLINICAL TRIAL: NCT06490315
Title: Effectiveness and Cost Effectiveness of a Mobile Psychoeducation Program (OkeyMind) for Social Anxiety Among Youth: A Randomized Controlled Trial
Brief Title: Effectiveness and Cost Effectiveness of OkeyMind for Social Anxiety Among Youth
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Shue Yan University (Other)
Responsible Party: Principal Investigator, Wang Yizhou, Assistant Professor, Hong Kong Shue Yan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OkeyMind intervention
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-03

CONDITIONS: Depression; Social Anxiety
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive a one-month mobile psychoeducation program (OkeyMind), which includes both psychoeducation and meditation components, with all content fully automated.
  Interventions: Behavioral: OkeyMind intervention
- Waiting list control group (Experimental): Participants in the waiting list control group will withhold access to the OkeyMind intervention until after the 3-month follow-up assessment.
  Interventions: Behavioral: Wait-list control

INTERVENTIONS:
Behavioral: OkeyMind intervention — The intervention group will receive a one-month mobile psychoeducation program (OkeyMind), which includes both psychoeducation and meditation components, with all content fully automated.
  Arms: Intervention group
Behavioral: Wait-list control — Participants in the waiting list control group will withhold access to the OkeyMind intervention until after the 3-month follow-up assessment.
  Arms: Waiting list control group

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness and cost-effectiveness of a mobile-based psychoeducation program (OkeyMind) in mitigating symptoms associated with social anxiety among youth.

Participants will be recruited and screened onsite and then randomized to the intervention group and the waiting list control group. The intervention group will receive a one-month mobile psychoeducation program (OkeyMind), which includes both psychoeducation and meditation components, with all content fully automated. The waiting list control group will receive the same intervention after 3 months. Participants will be followed up at three time-points: baseline, 1 month, and 3 months Results: The investigators will recruit 180 participants, with 90 in each group. The primary effectiveness outcomes are the scores of SPIN and PHQ-9, and the cost-effectiveness outcomes is measured by the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L).

This research evaluates the effectiveness and cost-effectiveness of OkeyMind, a mobile-based psychoeducation program for youth with social anxiety. OkeyMind might be a promising strategy for combating social anxiety, especially in low- and middle-income countries with limited medical resources. By leveraging mobile technology, it aims to provide accessible, cost-effective mental health support, improving outcomes on a broader scale.

DETAILED DESCRIPTION:
Background: Social anxiety is increasingly prevalent among youths, leading to social withdrawal and isolation, which heighten depression risk. eHealth interventions have shown promise in improving access and engagement, offering anonymity, broader accessibility, and personalized treatment features. However, the effectiveness and cost-effectiveness of eHealth methods for young individuals dealing with social anxiety-driven depression remain unexplored.

Objective: This randomized controlled trial aims to evaluate the effectiveness and cost-effectiveness of a mobile-based psychoeducation program (OkeyMind) in mitigating symptoms associated with social anxiety among youth.

Methods: Participants will be recruited and screened onsite and then randomized to the intervention group and the waiting list control group. Eligible participants are youths aged 18 to 25 years with moderate or above depression [Patient Health Questionnaire-9 (PHQ-9)>9), mild or above social phobia [Social Phobia Inventory (SPIN)>19], and a smartphone with WeChat installed. The intervention group will receive a one-month mobile psychoeducation program (OkeyMind), which includes both psychoeducation and meditation components, with all content fully automated. The waiting list control group will receive the same intervention after 3 months. Participants will be followed up at three time-points: baseline, 1 month, and 3 months Results: The investigators will recruit 180 participants, with 90 in each group. The primary effectiveness outcomes are the scores of SPIN and PHQ-9, and the cost-effectiveness outcomes is measured by the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L). Participant recruitment will begin before January 2025. The first follow-up assessment will conclude by May 2025, and data analysis will be finalized by early 2026. Results will be expected around May 2026.

Conclusions: This research evaluates the effectiveness and cost-effectiveness of OkeyMind, a mobile-based psychoeducation program for youth with social anxiety. OkeyMind might be a promising strategy for combating social anxiety, especially in low- and middle-income countries with limited medical resources. By leveraging mobile technology, it aims to provide accessible, cost-effective mental health support, improving outcomes on a broader scale.

ELIGIBILITY:
Inclusion Criteria:

1. youths aged between 15 and 24 years old;
2. exhibiting mild or above social phobia (i.e. Social Phobia Inventory score ≥ 25);
3. having a smartphone with WeChat installed and basic internet literacy

Exclusion Criteria:

1. unable to attempt a baseline assessment (e.g., due to being unpermitted to leave a psychiatric ward);
2. currently receiving another intensive psychological intervention;
3. currently holding active suicidal plan;
4. currently diagnosed with psychological disorders (e.g., schizophrenia, bipolar disorder, etc.).

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Social Phobia Inventory | 3 months
  Developed by Connor et al. in 2000, SPIN is a brief self-report tool consisting of 17 items that assess fear, avoidance, and physiological discomfort in social situations. It is specifically designed for use with social anxiety disorder. A cut-off value of 19 is used to distinguish between clients with and without social phobia.
Patient Health Questionnaire-9 | 3 months
  The Patient Health Questionnaire-9 (PHQ-9) is widely used to screen for the presence and severity of depression, monitor the severity of depression over time, and assist with the diagnosis of depression. Each of the nine items is scored from 0 (not at all) to 3 (nearly every day), with a total score ranging from 0 to 27. Higher scores indicate more severe depressive symptoms. PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.

SECONDARY OUTCOMES:
EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) | 3 months
  EQ-5D-5L is an established tool for assessing the general health status of individuals across a wide array of health conditions and treatments. It measures health outcomes in five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a five-level scale, from no problems (level 1) to extreme problems (level 5), facilitating a comprehensive evaluation of a patient's health-related quality of life. The total score is derived by converting the individual dimension scores into a single summary index value, reflecting the overall health status, with higher scores indicating better health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhou Wang, PhD, Principal Investigator — Hong Kong Shue Yan University
Locations (1):
- Hong Kong Shue Yan University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang YZ, Zhou DR, Ng SM, Wang BB, Feng YY, Weng X. Effectiveness and Cost-Effectiveness of a Mobile Psychoeducation Program (OkeyMind) for Social Anxiety Symptoms Among Youths: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jul 14;14:e64518. doi: 10.2196/64518. PMID 40658950